CLINICAL TRIAL: NCT00597766
Title: Clinical Trials in Stroke Rehabilitation
Brief Title: Subacromial Corticosteroid Injection for Hemiplegic Shoulder Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, John Chae, MD, Prof Vice Chair Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K24HD054600 (NIH); K24HD054600 (NIH)
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Shoulder Pain
Keywords: CVA; Hemiplegia; Hemiplegic shoulder pain; Subacromial steroid injection
MeSH Terms: conditions — Shoulder Pain; Hemiplegia | interventions — Lidocaine; Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Active Comparator): Drug: Lidocaine (Neer's Test)
  Drug: 20 mg Triamcinolone + Lidocaine
  Interventions: Drug: Lidocaine; Drug: Triamcinolone + Lidocaine
- Standard Dose (Active Comparator): Drug: Lidocaine (Neer's Test)
  Drug: 40 mg Triamcinolone + Lidocaine
  Interventions: Drug: Lidocaine; Drug: Triamcinolone + Lidocaine
- High Dose (Experimental): Drug: Lidocaine (Neer's Test)
  Drug: 60 mg Triamcinolone + Lidocaine
  Interventions: Drug: Lidocaine; Drug: Triamcinolone + Lidocaine

INTERVENTIONS:
Drug: Lidocaine — One-time Screening/Eligibility Neer's Test: 5 cc of 2% lidocaine
Drug: Triamcinolone + Lidocaine — Low Dose -- One-time injection of 20 mg triamcinolone: 1.5 cc of normal saline, 0.5 cc of 40mg/cc of triamcinolone and 2 cc of 2% lidocaine
  Other Names: Kenalog = Triamcinolone
  Arms: Low Dose
Drug: Triamcinolone + Lidocaine — Standard Dose -- One-time injection of 40 mg triamcinolone: 1 cc of normal saline, 1 cc of 40mg/cc of triamcinolone and 2 cc of 2% lidocaine
  Other Names: Kenalog = Triamcinolone
  Arms: Standard Dose
Drug: Triamcinolone + Lidocaine — High Dose -- One-time injection of 60 mg triamcinolone: 0.5 cc of normal saline, 1.5 cc of 40mg/cc of triamcinolone and 2 cc of 2% lidocaine
  Other Names: Kenalog = Triamcinolone
  Arms: High Dose

SUMMARY:
This is a double-blinded study of subacromial corticosteroid injection (steroid injection to the shoulder) to treat shoulder pain in the paralyzed (hemiplegic) shoulder of chronic stroke survivors. This study is designed to evaluate pain relief of a standard steroid injection treatment, compared to a high dose treatment and a low dose treatment, for shoulder pain in stroke survivors. A total of 105 chronic stroke survivors with moderate to severe shoulder pain will be enrolled. All eligible participants will undergo an initial test injection to localize pain to the subacromial space. If this turns out to be positive, the subjects will be randomly assigned to one of three groups:

1. low dose group which receives 20mg of steroid (triamcinolone) injection to the subacromial space of the affected shoulder;
2. standard dose group which receives a standard 40mg of steroid (triamcinolone) injection to the subacromial space of the affected shoulder; or
3. high dose group which receives 60mg of steroid (triamcinolone) injection to the subacromial space of the affected shoulder.

Study participants will all rate their pain in interviews (Baseline, weeks 1, 2, 3, 4, 8, 12 (7 times) and in laboratory-based measures that will be administered at baseline, weeks 4, 8, 12 (4 times). Subjects will be followed for a total of 13 weeks.

The study will thus characterize the dose response of triamcinolone for the treatment of hemiplegic shoulder pain.

DETAILED DESCRIPTION:
* A total of 105 chronic stroke survivors with moderate to severe shoulder pain will be enrolled. Subjects will be enrolled in the study for 13 weeks. Subjects who complete the protocol will visit MetroHealth five times.
* Visit 1: Baseline information about demographics, past medical history, and inclusion/exclusion issues will be collected for study participants. Pertinent lab work will be performed to determine initial eligibility.
* Visit 2: All initially eligible participants also will undergo a test injection of lidocaine to localize the pain to the subacromial bursa (Neer's Test). A positive Neer's test is required to finalize eligibility for further participation. Participants who satisfy inclusion/exclusion criteria (including a positive Neer's test) will be randomized to high dose steroid, standard dose steroid, or low dose steroid via a computer generated random number table. The study participants and the observer will be blinded as to these groupings.
* After the initial Neer's test and randomization, participants will receive their assigned injection the same day. Participants then will be followed for an additional 12 weeks, including three follow-up visits (Visits 3-5). The total participation time in this study will be 13 weeks.
* The primary outcome measure will be the BPI 12. The BPI is a pain questionnaire, which assesses the "worst pain" in the previous 7 days. Secondary outcome measures also will be assessed together with BPI 12. There will be 3 additional secondary outcome measures, Fugl-Meyer Motor Assessment (a measure of poststroke motor impairment), pain free external rotation range of motion (ROM) and pain free abduction ROM.
* A blinded therapist will administer all outcome measures. The primary outcome will be assessed on a weekly basis via telephone (or in person during weeks of MetroHealth visits) starting on the day of Visit 1 and continuing to 12-weeks after steroid injection (i.e., for the 13 weeks of the subject's participation). The remaining secondary outcomes will be assessed in clinic visits at least every 4 weeks starting with Visit 2 (Visits 2-5).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* upper extremity hemiplegia due to hemorrhagic or nonhemorrhagic stroke
* ≤ 4/5 on manual muscle testing for the deltoid on the affected side if isolated movement is present
* post-stroke duration ≥ 1-mo, but < 24-mo
* shoulder pain sustained for ≥ 1-mo
* BPI 12 ≥ 4 (pain scale)
* willing and able to report pain and other conditions throughout the 4-mo study period
* positive Neer's test

Exclusion Criteria:

* evidence of joint or overlying skin infection
* > 2 opioid and/or nonopioid analgesic for shoulder pain (i.e., > 2 regardless of class)
* regular intake of pain medications for any other chronic pain
* steroid injections to the shoulder in the last 6-wks
* history of pre-stroke shoulder pain
* bleeding disorder
* for those on Coumadin, INR > 3.0
* history of allergies to lidocaine
* renal insufficiency (Creat > 2.0)
* both history of liver disease & abnormal liver enzyme lab results
* poorly controlled diabetes (HbA1c > 7.0)
* medical instability
* cognitive deficits; In order to pass the cognitive exam, the participant must exhibit 3/3 registration and recall the same three objects in 30 minutes. The participant must also be able to correctly rank the following three levels of pain from highest to lowest: 1) falling from a 2-story building and breaking both ankles, 2) stubbing one's toe and 3) getting bitten by a mosquito.
* immunocompromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Chae, MD, Principal Investigator — MetroHealth Medical Center; Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org/body.cfm?id=2438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from an urban, academic rehabilitation center from 10/2007 to 6/2012 in the United States.
Pre-assignment Details: Subjects had to have a positive Neer's test (50% pain reduction by subacromial lidocaine) to be enrolled and randomized. 59 were screened. 28 subjects were consented and enrolled.
Groups:
- 20mg Triamcinolone: Low dose group.
- 40mg Triamcinolone: Standard dose group
- 60mg Triamcinolone: High dose group
Period: Enrolled
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Started | 9 | 9 | 10
Completed | 9 | 9 | 10
Not Completed | 0 | 0 | 0
Period: Follow-up 1, Week 4
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Started | 9 | 9 | 10
Completed | 8 | 9 | 10
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Follow-up 2, Week 8
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Started | 8 | 9 | 10
Completed | 8 | 9 | 9
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Follow-up 3, Week 12
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Started | 8 | 9 | 9
Completed | 8 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants was determined on a power analysis. The goal was 31 subjects per group.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone | Total
Number analyzed (Participants) | 9 | 9 | 10 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 9 | 24
  >=65 years | 2 | 1 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (7.1) | 54.7 (10.2) | 54.0 (9.9) | 55.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 5 | 6 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: BPI 12 (Brief Pain Inventory, Question 12) Pain Questionnaire
Description: Change in BPI-12, Worst pain in the last week on 0 (No Pain) to 10 (Worst Pain Possible) scale, from baseline to week 12. The data in the Outcome Measure data table represent the comparison of week 12 to baseline using least squares means from the linear mixed model, but data from all time points are included in the Statistical Analyses to arrive at the reported slopes/group x time interactions.
Time Frame: Baseline, weeks 1, 2, 3, 4, 8, 12 (7 times)
Population: We used available-cases. Missing values handled with maximum likelihood methods.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Number analyzed (Participants) | 9 | 9 | 10
units on a scale | -1.7 [-3.9 to 0.6] | -2.2 [-4.4 to 0.0] | -4.7 [-6.8 to -2.5]
Statistical Analysis 1: Comparison: 20mg Triamcinolone vs 60mg Triamcinolone; Hypothesis that 60mg group would have greater pain relief than the the 20mg group. The study was powered to detect the difference in pain between the 40mg and placebo at 4-wks. To detect effect size 0.75 with alpha of 0.05, beta of 0.20, 31 the difference between the 60mg and placebo groups (effect size > 1.0),18 participants per group are needed. *NOTE* the design was changed from placebo-control due to ethical concerns arising from ethical concerns of placebo injection; Test type: Superiority or Other; p = 0.16, Linear mixed model — Comparison 60mg vs. 20mg: F (1,92)=2.06, p=0.16; 1st order antedependence covariance structure; GroupXtime interaction = -0.17
Statistical Analysis 2: Comparison: 20mg Triamcinolone vs 40mg Triamcinolone; Hypothesis that 40mg group would have greater pain reduction than the 20mg group. The study was powered to detect the difference in pain between the 40mg and placebo at 4-wks. To detect effect size 0.75 with alpha of 0.05, beta of 0.20, 31 the difference between the 60mg and placebo groups (effect size > 1.0),18 participants per group are needed. *NOTE* the design was changed from placebo-control due to ethical concerns arising from ethical concerns of placebo injection; Test type: Superiority or Other; p = 0.77, linear mixed model — Comparison 40mg vs. 20mg: F (1,90)=0.1, p=0.77; first order antedependent covariance structure; group x time interaction = -0.04

2. Secondary Outcome: Fugl-Meyer Motor Assessment, Upper Limb Domain
Description: Evaluates and measures recovery in post-stroke hemiplegic patients. Items are scored on a 3-point ordinal scale:
  0 = cannot perform
  1. = performs partially
  2. = performs fully Scores for 33 motor function items are summed to arrive at a total score ranging from 0 to 66, where higher scores indicate greater motor function Differences baseline to week 12. The data in the Outcome Measure data table represent the comparison of week 12 to baseline using least squares means from the linear mixed model, but data from all time points are included in the Statistical Analyses to arrive at the reported slopes/group x time interactions.
Time Frame: Baseline, weeks 4, 8, 12 (4 times)
Population: Available-case analysis with missing data handled by maximum likelihood methods.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Number analyzed (Participants) | 9 | 9 | 10
units on a scale | 5.1 [-0.1 to 10.4] | 4.5 [-0.9 to 9.8] | 2.3 [-2.8 to 7.4]
Statistical Analysis 1: Comparison: 20mg Triamcinolone vs 60mg Triamcinolone; This study was not powered for secondary outcomes. The effect of treatment group over time was analyzed using a linear mixed model for repeated measures with random intercept and subject effects. The dependent variable was treatment group and variables for week (continuous) and group interaction term was included in the model. The effect of treatment at discrete time points was analyzed using a linear mixed model with categorical time; Test type: Superiority or Other; p = 0.2, Linear mixed model — Comparison 60mg vs. 20mg: F (1,36)=1.7, p=0.2; first order antedpendent covariance structure; group x time interaction = -0.3
Statistical Analysis 2: Comparison: 20mg Triamcinolone vs 40mg Triamcinolone; This study was not powered for secondary outcomes.The effect of treatment group over time was analyzed using a linear mixed model for repeated measures with random intercept and subject effects. The dependent variable was treatment group and variables for week (continuous) and group interaction term was included in the model. The effect of treatment at discrete time points was analyzed using a linear mixed model with categorical time; Test type: Superiority or Other; p = 0.9, linear mixed model — Comparison 40mg vs. 20mg: F (1,35)=0.0, p=0.9; 1st order antedependence covariance structure; group x time interaction = -0.02

3. Secondary Outcome: Pain Free External Rotation Range of Motion (ROM)
Description: Differences in least-mean squares (Degrees) from baseline to week 12. The data in the Outcome Measure data table represent the comparison of week 12 to baseline using least squares means from the linear mixed model, but data from all time points are included in the Statistical Analyses to arrive at the reported slopes/group x time interactions.
Time Frame: Baseline, weeks 4, 8, 12 (4 times)
Population: Available-case analysis with missing data handled by maximum likelihood methods.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Number analyzed (Participants) | 9 | 9 | 10
units on a scale | 26.7 [8.2 to 45.1] | 12.7 [-6.0 to 31.4] | 10.3 [-7.5 to 28.1]
Statistical Analysis 1: Comparison: 20mg Triamcinolone vs 60mg Triamcinolone; The study was not powered for secondary analyses. The effect of treatment group over time was analyzed using a linear mixed model for repeated measures with random intercept and subject effects. The dependent variable was treatment group and variables for week (continuous) and group interaction term was included in the model. The effect of treatment at discrete time points was analyzed using a linear mixed model with categorical time; Test type: Superiority or Other; p = 0.2, linear mixed model — Comparison 60mg vs. 20mg: F (1,36)=1.6, p=0.2; unstructured covariance structure; Groupxtime interaction = 1.3
Statistical Analysis 2: Comparison: 20mg Triamcinolone vs 40mg Triamcinolone; Secondary outcomes were not powered for analysis. The effect of treatment group over time was analyzed using a linear mixed model for repeated measures with random intercept and subject effects. The dependent variable was treatment group and variables for week (continuous) and group interaction term was included in the model. The effect of treatment at discrete time points was analyzed using a linear mixed model with categorical time; Test type: Superiority or Other; p = 0.3, linear mixed model — Comparison 40mg vs. 20mg: F (1,35)=1.0, p=0.3; Unstructured covariance structure; Groupxtime interaction = 1.1

4. Secondary Outcome: Pain Free Abduction Range of Motion (ROM)
Description: Difference in least-squares means (Degrees) from baseline to week 12. The data in the Outcome Measure data table represent the comparison of week 12 to baseline using least squares means from the linear mixed model, but data from all time points are included in the Statistical Analyses to arrive at the reported slopes/group x time interactions.
Time Frame: Baseline, weeks 4, 8, 12 (4 times)
Population: Available-case analysis with missing data handled by maximum likelihood methods.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Number analyzed (Participants) | 9 | 9 | 10
units on a scale | 33.3 [7.9 to 58.7] | 15.2 [-10.6 to 41.0] | 28.0 [3.3 to 52.6]
Statistical Analysis 1: Comparison: 20mg Triamcinolone vs 60mg Triamcinolone; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.8, linear mixed model — Comparison 60mg vs. 20mg: F (1,36)=0.06, p=0.8; first order antedepentent covariance structure; group x time interaction = 0.4
Statistical Analysis 2: Comparison: 20mg Triamcinolone vs 40mg Triamcinolone; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.3, linear mixed model — Comparison 40mg vs. 20mg: F (1,35)=1.1, p=0.3; first order antedependent covariance structure; group x time interaction = 1.7

ADVERSE EVENTS:
Arm/Group | 20mg Triamcinolone | 40mg Triamcinolone | 60mg Triamcinolone
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 1/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20mg Triamcinolone (N=9) | 40mg Triamcinolone (N=9) | 60mg Triamcinolone (N=10)
GI Illness requiring hospitalization (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Subject hospitalized for gastrointestinal illness. Unrelated to study.

LIMITATIONS AND CAVEATS:
The study was powered to detect differnces between high-dose and placebo, and standard-dose and placebo. The trial was altered due to ethical concerns for placebo injection due to apparent effectiveness in the literature. Low dose was substituted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No